CLINICAL TRIAL: NCT02719899
Title: Pilot Study to Evaluate the Effect of Fasting and Refeeding on T-Cell Fate
Brief Title: Effect of Fasting and Refeeding on T-cell Fate
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160085; 16-H-0085
Record Dates: First submitted 2016-03-24; First posted 2016-03-25 (Estimated); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Asthma; Inflammation
Keywords: NLRP3 Inflammasome; Sirtuin 3; T-Cell Polarity; Caloric Restriction; Natural History
MeSH Terms: conditions — Asthma; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Healthy Volunteers

SUMMARY:
Background:

Researchers want to better understand the body s immune response to calorie restriction. To do this, they are asking healthy volunteers to fast for 24 hours. Researchers will test immune response before and after fasting.

Objectives:

To explore the benefits of calorie restriction on immune health.

Eligibility:

Healthy volunteers ages 21 to 37 with a body mass index between 22 and 29.

Design:

Participants will be screened with medical history, physical exam, and blood tests.

Participants will visit NIH after an overnight fast. Their baseline immune response will be taken. They will give blood and urine samples. Then they will be given breakfast. This visit will take about 2 hours.

Participants will fast (not eat or drink anything except water) for the next 24 hours. They will return to NIH the next morning. Their immune response will be taken. They will give blood and urine samples. Then they will be given breakfast. Their immune response will be taken 3 hours later. They will give a blood sample. This visit will take about 4 hours.

DETAILED DESCRIPTION:
Intermittent caloric restricted or fasting has numerous health effects including the reduction in numerous cardiovascular and pulmonary disease risk factors. The cellular programs activated by caloric restriction are similarly regulated in preclinical and clinical studies in response to a 24-hour fast. We have found that a beneficial effect of a 24-hour fasting blunts the activation of a component of the innate immune system, termed the NLRP3 inflammasome. This inflammasome, as a mediator of sterile inflammation, is associated with the development of diabetes, asthma and atherosclerosis. At the same time, we found that refeeding after the 24-hour fast significantly increased NLRP3 protein levels. As NLRP3 is increased in obesity, the nutrient intervention (24 hour fast and then refeeding) we studied may be useful to evaluate nutrient-overload effects on the immune system. Pertaining to this it has recently been found in a preclinical study that NLRP3 can also orchestrate differentiation of na(SqrRoot) ve T cells into T(H)2 cells. Interestingly both the NLRP3 inflammasome and T(H)2 cell activation contribute to asthma. In this context we hypothesize that the assessment of the effect on refeeding on T(H)2 cell differentiation (polarity) may allow us to dissect out the mechanisms underpinning nutrient overload induced T(H)2 cell activation. To evaluate this blood samples to test T-cell biology will be collected in subjects, at baseline, after a fixed caloric meal and in response to a 24-hour fast (water intake will not be restricted). The objective of this pilot study is to identify if nutrient-load regulates T-Cell differentiation capacity and to test whether this pathway could be investigated as a therapeutic target to blunt/negate the inflammation associated with nutrient-excess associated diseases including asthma.

ELIGIBILITY:
* INCLUSION CRITERIA:

As this is a pilot study, the age-range and BMI range of subjects will be restricted to potentially reduce metabolic variables associated with a wide age- and BMI-range.

* Males and females between the ages of 21 and 37
* BMI greater than or equal to 22 and less than 30

EXCLUSION CRITERIA:

* Subjects with an acute or chronic illness as per history, on laboratory analysis or due to use of medications
* Subjects taking vitamins or supplements or any medications, except oral contraceptives, within 4 weeks of participation into this study
* BMI less than 22 or greater than or equal to 30
* Female subjects who are pregnant or lactating
* Subjects who have donated blood or participated in another clinical trial involving blood draws in the last 8 weeks
* Subjects who use nicotine products

Ages: 21 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: -Males and females between the ages of 21 and 37 @@@-BMI greater than or equal to 22 and less than 30
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-02-24 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the change in TH2 cell cytokine (IL-4, IL-5 and/or IL-13) secretion in response to T-cell differentiation comparing the fasted to the refeeding response. | 24 hours
  The comparisons will be performed using paired two-tailed Student t-tests. Significance will be tested at the 0.05 alpha level in this pilot study

SECONDARY OUTCOMES:
To identify if nutrient-load regulates T-Cell differentiation capacity and to test whether this pathway could be investigated as atherapeutic target to blunt/negate the inflammation associated with nutrient-excess associated diseases includin... | Visit 3, 3hrs post-meal
  Blood samples to test T-cell biology will be collected in subjects, at baseline, after a fixed caloric meal and in response to a 24-hour fast (water intake will not be restricted). Analysis of T-cell interleukin expression and regulation and mitochondrial functioning in primary T-cells. Analysis of mitochondrial biology in these immune-modulatory effects.
Evaluate whether these effects are associated with activation of the Sirt3 and its canonical mitochondrial adaptive programs. | Visit 3, 3hrs post-meal
  Analysis of difference in additional T-cell polarity signatures. Analysis ofcytokine and other protein levels in serum comparing the fed versus fasted states. Analysis of serum metabolites that may be modulating T-cell polarity.

CONTACTS AND LOCATIONS:
Overall Officials: Michael N Sack, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sack MN, Finkel T. Mitochondrial metabolism, sirtuins, and aging. Cold Spring Harb Perspect Biol. 2012 Dec 1;4(12):a013102. doi: 10.1101/cshperspect.a013102. PMID 23209156
- [Background] Fontana L, Meyer TE, Klein S, Holloszy JO. Long-term calorie restriction is highly effective in reducing the risk for atherosclerosis in humans. Proc Natl Acad Sci U S A. 2004 Apr 27;101(17):6659-63. doi: 10.1073/pnas.0308291101. Epub 2004 Apr 19. PMID 15096581
- [Background] Fontana L, Partridge L. Promoting health and longevity through diet: from model organisms to humans. Cell. 2015 Mar 26;161(1):106-118. doi: 10.1016/j.cell.2015.02.020. PMID 25815989
- [Derived] Han K, Singh K, Rodman MJ, Hassanzadeh S, Wu K, Nguyen A, Huffstutler RD, Seifuddin F, Dagur PK, Saxena A, McCoy JP, Chen J, Biancotto A, Stagliano KER, Teague HL, Mehta NN, Pirooznia M, Sack MN. Fasting-induced FOXO4 blunts human CD4+ T helper cell responsiveness. Nat Metab. 2021 Mar;3(3):318-326. doi: 10.1038/s42255-021-00356-0. Epub 2021 Mar 15. PMID 33723462
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-H-0085.html